CLINICAL TRIAL: NCT02093416
Title: Leptin Receptors in the Bariatric Surgical Population Within the University of Pittsburgh Medical System: A Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO13010529
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Obesity; Leptin
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: Control Group: BMI <30 There are 20 controls in this group
- Group 2: BMI 30-35 There were 12 controls in this class
- Group 3: BMI 35-40 There were 9 controls in this clas
- Group 4: BMI >40 There were 9 controls in this class

SUMMARY:
Prospective cohort study evaluating the role of leptin receptors in the bariatric surgical population compared with non obese controls. Additionally serum levels of leptin, ghrelin, motilin and PYY will be compared amongst the different BMI classes and a quality of life questionnaire completed by all participants.

The hypothesis is that obese individuals have lower leptin receptors in enterocytes which is partially responsible for the higher serum leptin levels without appropriate control of satiety.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic Intervention

Exclusion Criteria:

* 18 years of age or older
* No acute GI bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and Females undergoing endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
PCR test for Leptin Receptors | 1 week
  Endoscopic biopsies of enterocytes will be measured via PCR

SECONDARY OUTCOMES:
ELISA test for ghrelin, motilin, leptin and PYY | 1 week
  Blood samples collected to determine hormones via ELISA
IWQOL lite questionnaire | 1 week
  Quality of Life questionnaire on obesity

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Seminerio, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh/UPMC Presby, Pittsburgh, Pennsylvania, United States